CLINICAL TRIAL: NCT07275996
Title: Effects of Creatine Monohydrate and β-Hydroxy-β-Methylbutyrate Supplementation Combined With Multicomponent Exercise on Physical Performance, Cognition and Quality of Life in Institutionalized Older Adults: A Randomized Double-Blind Parallel-Group Trial
Brief Title: Neuromuscular and Multi-Omics Synergy of Combined Creatine × HMB Supplementation Plus Exercise to Improve Muscle Function in Sarcopenic Frailty
Acronym: MULTI-FRAIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Principal Investigator, Juan Francisco Mielgo, Full Professor of Physiology, Principal Investigator, Universidad de Burgos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBU-FB-CREHMB-CRXO-2025; IR 24/2023 (Other: Ethics Committee Approval Number)
Record Dates: First submitted 2025-09-29; First posted 2025-12-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Frailty; Sarcopenia; Aging; Malnutrition Elderly
Keywords: creatine; HMB; supplementation; multicomponent exercise; concurrent training; institutionalized older adults; nursing home; physical performance; quality of life; oxidative stress; inflammation; geriatric assessment; multi-omics; microRNA; proteomics
MeSH Terms: conditions — Frailty; Sarcopenia; Inflammation | interventions — Cellulose; Creatine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group clinical trial with four study arms. Participants will receive 12 weeks of dietary supplementation combined with a supervised multicomponent exercise program, followed by a 3-month follow-up period without supplementation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blind design: Participants, care providers (exercise supervisors and supplement distributors), investigators, and outcome assessors will remain blinded to allocation. Supplements will be provided in identical sachets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Creatine + HMB + Exercise (Experimental): Participants receive a total of 6 g/day of powder consisting of 3 g/day of creatine monohydrate and 3 g/day of β-hydroxy-β-methylbutyrate (HMB), administered once daily, combined with a supervised multicomponent exercise program for 12 weeks.
  Interventions: Dietary Supplement: Creatine Monohydrate; Behavioral: Multicomponent Exercise Program; Dietary Supplement: β-Hydroxy-β-Methylbutyrate (HMB)
- Placebo + Exercise (Placebo Comparator): Participants receive a total of 6 g/day of cellulose (placebo), administered once daily, combined with a supervised multicomponent exercise program for 12 weeks.
  Interventions: Dietary Supplement: Placebo (Cellulose); Behavioral: Multicomponent Exercise Program
- Creatine + Exercise (Active Comparator): Participants receive a total of 6 g/day of powder consisting of 3 g/day of creatine monohydrate and 3 g/day of cellulose (placebo filler), administered once daily, combined with a supervised multicomponent exercise program for 12 weeks.
  Interventions: Dietary Supplement: Placebo (Cellulose); Dietary Supplement: Creatine Monohydrate; Behavioral: Multicomponent Exercise Program
- HMB + Exercise (Active Comparator): Participants receive a total of 6 g/day of powder consisting of 3 g/day of β-hydroxy-β-methylbutyrate (HMB) and 3 g/day of cellulose (placebo filler), administered once daily, combined with a supervised multicomponent exercise program for 12 weeks.
  Interventions: Dietary Supplement: Placebo (Cellulose); Behavioral: Multicomponent Exercise Program; Dietary Supplement: β-Hydroxy-β-Methylbutyrate (HMB)

INTERVENTIONS:
Dietary Supplement: Placebo (Cellulose) — Sachets containing cellulose used as placebo filler to match supplement volume, appearance, and taste. Administered once daily, mixed with yogurt or juice, during the intervention period.
  Arms: Creatine + Exercise; HMB + Exercise; Placebo + Exercise
Dietary Supplement: Creatine Monohydrate — Sachets containing creatine monohydrate used as an active dietary supplement. Administered once daily during the intervention period.
  Arms: Creatine + Exercise; Creatine + HMB + Exercise
Behavioral: Multicomponent Exercise Program — Supervised exercise sessions, 4 times per week (~60 minutes each), including resistance, endurance, balance, coordination, and flexibility training. Intensity adapted to participants' functional status (Borg scale 6-9). Conducted throughout the 12-week intervention period.
Dietary Supplement: β-Hydroxy-β-Methylbutyrate (HMB) — Sachets containing calcium β-hydroxy-β-methylbutyrate used as an active dietary supplement. Administered once daily during the intervention period.
  Arms: Creatine + HMB + Exercise; HMB + Exercise

SUMMARY:
Sarcopenia and physical frailty are highly prevalent among institutionalized older adults and are major contributors to functional decline, reduced mobility, and loss of independence. Combined exercise and targeted nutritional strategies have emerged as promising approaches to mitigate these age-related impairments.

This randomized, double-blind, placebo-controlled, parallel-group clinical trial aims to evaluate the independent and combined effects of creatine monohydrate (CRE) and β-hydroxy-β-methylbutyrate (HMB), administered alongside a supervised multicomponent exercise program, on physical function, body composition, cognitive performance, and quality of life in institutionalized older adults with physical frailty and sarcopenia.

A total of 80 adults aged ≥65 years will be randomized to one of four intervention groups for 12 weeks: placebo plus exercise, creatine plus exercise, HMB plus exercise, or creatine plus HMB plus exercise. A supplement-free follow-up period will be conducted to evaluate the sustainability of intervention effects.

In addition to clinical and functional outcomes, the study incorporates molecular and biological assessments to explore mechanistic pathways underlying functional adaptation and interindividual variability in response to the interventions.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel-group clinical trial is designed to evaluate the independent and combined effects of creatine monohydrate (CRE) and β-hydroxy-β-methylbutyrate (HMB) supplementation when administered alongside a structured multicomponent exercise program in institutionalized older adults with physical frailty and sarcopenia. Sarcopenia and frailty are highly prevalent in this population and are associated with functional disability, increased health care utilization, and reduced quality of life. Nutritional strategies targeting muscle metabolism, when combined with systematic exercise, may attenuate functional decline and improve health outcomes in this vulnerable group.

Study Population and Design

A total of 80 institutionalized adults aged ≥65 years will be recruited from nursing homes in the province of Burgos (Spain). Participants will be stratified by sex and randomized to one of four parallel intervention groups for a 12-week intervention period: placebo plus exercise, creatine plus exercise, HMB plus exercise, or creatine plus HMB plus exercise. All intervention groups will be followed by a supplement-free follow-up period to assess the persistence of intervention effects.

Intervention

Dietary supplementation will be administered once daily using identical sachets to ensure blinding and equivalent supplement volume across groups. Participants will receive a total of 6 g/day of powder, consisting of cellulose (placebo), creatine monohydrate, HMB, or their combinations, depending on group allocation. Supplement administration will be supervised by nursing staff and mixed with food or beverages according to standard procedures.

All participants will complete a supervised multicomponent exercise program conducted four times per week (~60 minutes per session). Exercise sessions will include resistance, balance, coordination, and flexibility training, with intensity individually adapted according to functional capacity using the Borg Rating of Perceived Exertion Scale.

Outcomes and Assessments

Clinical, functional, cognitive, and quality-of-life assessments will be conducted at baseline, post-intervention (Week 12), and during follow-up. Primary and secondary outcome measures focus on physical performance, muscle strength, body composition, cognitive function, activities of daily living, nutritional status, and quality of life.

Molecular and Biological Assessments

In addition to clinical outcomes, the study incorporates biological and molecular assessments to explore mechanistic pathways underlying functional adaptation and interindividual variability in response to supplementation and exercise. Venous blood samples will be collected for the analysis of inflammatory markers, oxidative stress and antioxidant status, hormonal profiles, and circulating and exosomal molecular signatures related to muscle metabolism and neuromuscular function. Body composition parameters will be assessed using dual-energy X-ray absorptiometry (DXA).

Statistical Analysis

Statistical analyses will be conducted using mixed-effects models appropriate for parallel-group randomized designs, with treatment group, time, and their interaction as fixed effects, and sex and age included as covariates where appropriate. Post-hoc pairwise comparisons will be adjusted for multiple testing. Statistical significance will be set at p < 0.05.

Ethics and Data Protection

The study was approved by the Ethics Committee of the University of Burgos (IR 24/2023). Written informed consent will be obtained from all participants or their legal representatives. All data will be pseudonymized and managed in accordance with the General Data Protection Regulation (GDPR) and Spanish data protection laws.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized older adults (≥65 years) residing in the Fuentes Blancas Nursing Home (Diputación de Burgos).
* Clinical diagnosis of frailty or sarcopenia according to validated criteria (e.g., Fried phenotype, SPPB ≤ 9, or low ALMI by DEXA).
* Ability to participate in an exercise program as assessed by the medical staff.
* Written informed consent provided by the participant or, if cognitively impaired, by a legally authorized representative.

Exclusion Criteria:

* Severe renal insufficiency (eGFR < 30 mL/min/1.73m²) or liver failure.
* Advanced heart failure (NYHA class III-IV) or unstable cardiovascular disease.
* Active cancer or other severe medical conditions that contraindicate participation.
* Severe cognitive impairment (MMSE < 10) precluding adherence to the program without caregiver support.
* Known allergy or intolerance to creatine, HMB, or inulin.
* Participation in another clinical trial within the past 3 months.
* Any condition that, in the opinion of the medical team, may compromise safety or adherence to the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, Week 12 (end of intervention), and 3-month follow-up
  The SPPB assesses lower-extremity physical function through balance, gait speed, and chair stand components, generating a total score ranging from 0 to 12 (higher scores indicate better physical performance). Only the total score will be analyzed as the primary outcome.
Timed Up and Go (TUG) | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Time in seconds to rise from a chair, walk 3 meters, turn around, return, and sit down. Lower times indicate better mobility and balance.
Appendicular Lean Mass (ALM, kg) by DEXA | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Appendicular lean mass (sum of arms and legs lean tissue) measured in kilograms using DEXA. Higher values indicate greater muscle mass in limbs.

SECONDARY OUTCOMES:
Grip Strength | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Maximal isometric handgrip strength measured in kilograms using a validated hydraulic dynamometer (e.g., Jamar Plus+). Each test performed with the dominant hand in seated position, elbow at 90°. Best of three attempts recorded.
Leg and Back Isometric Strength | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Maximal isometric strength of leg and back extensors assessed in kilograms using a back/leg dynamometer (e.g., Baseline Evaluation Dynamometer). Participants stand on the platform and pull a fixed bar upwards. Best of two attempts recorded.
Seated Arm Curl Test | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Dynamic strength/endurance of upper limbs measured as the number of full arm curl repetitions in 30 seconds using a 2 kg dumbbell for women and a 4 kg dumbbell for men. Participants are seated upright without armrests.
Barthel Index | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Measure of independence in activities of daily living (feeding, bathing, mobility, toileting, etc.). Score ranges from 0 (total dependence) to 100 (independent).
Mini Nutritional Assessment (MNA) | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Validated tool to screen and assess nutritional status in older adults. Score ranges from 0-30 (higher = better nutritional status).
Cognitive Function - Mini-Mental State Examination (MMSE) | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Cognitive function assessed using the Mini-Mental State Examination (MMSE). Scores range from 0 to 30, with higher scores indicating better cognition.
Quality of Life - World Health Organization Quality of Life-Brief (WHOQOL-BREF) | Baseline, Week 12 (end of intervention), and 3-month follow-up
  26-item validated questionnaire covering physical, psychological, social and environmental domains.
  Scores range from 26 to 130; higher scores indicate better perceived quality of life.
Total Lean Mass (kg) by DEXA | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Whole-body lean soft tissue mass measured in kilograms using DEXA (Hologic Discovery or GE Lunar system) with manufacturer's software and standardized positioning. Higher values indicate greater muscle mass.
Total Fat Mass (percent body weight) by DEXA | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Whole-body fat mass measured with DEXA and expressed as a percentage of total body weight. Higher values indicate greater adiposity.
Visceral Adipose Tissue (VAT, cm³) by DEXA | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Visceral adipose tissue (VAT) volume estimated by DEXA in the android region of interest, expressed in cubic centimeters (cm³). Higher values indicate greater central adiposity.
Whole-Body Bone Mineral Density (BMD, g/cm²) by DEXA | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Whole-body BMD measured by DEXA, expressed as grams per square centimeter (g/cm²). Higher values indicate greater bone mineral density.
Cognitive Function - MEC (Spanish Adaptation of MMSE) | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Cognitive function assessed using the MEC (Spanish version of the MMSE). Scores range from 0 to 35, with higher scores indicating better cognition.
Number of Falls | Baseline to 3-month follow-up
  Incidence of falls recorded by nursing staff during the study period. Unit: number of events per participant. Lower numbers indicate better outcomes.
Number of Hospitalizations | Baseline to 3-month follow-up
  Incidence of hospital admissions for any cause. Unit: number of events per participant. Lower numbers indicate better outcomes.
Incidence of Respiratory and Urinary Infections | Baseline to 3-month follow-up
  Number of documented respiratory and/or urinary tract infections. Unit: number of events per participant. Lower numbers indicate better outcomes.
Incidence of Pressure Ulcers | Baseline to 3-month follow-up
  Number of new pressure ulcers recorded by nursing staff. Lower numbers indicate better outcomes.
Incidence of Urinary or Fecal Incontinence | Baseline to 3-month follow-up
  Occurrence of urinary and/or fecal incontinence episodes recorded in clinical charts. Lower numbers indicate better outcomes.
Serum C-reactive protein (CRP, mg/L) | Baseline, Week 12 (end of intervention)
  CRP will be measured in serum samples using a high-sensitivity ELISA. Results expressed in mg/L. Higher values indicate greater systemic inflammation.
Interleukin-6 (IL-6, pg/mL) | Baseline, Week 12 (end of intervention)
  Serum IL-6 concentration will be measured by ELISA and expressed in pg/mL. Higher values indicate greater systemic inflammation.
Tumor Necrosis Factor-alpha (TNF-α, pg/mL) | Baseline, Week 12 (end of intervention)
  Serum TNF-α concentration will be determined by ELISA and expressed in pg/mL. Higher values indicate greater systemic inflammation.
Reduced Glutathione (GSH, µmol/L) | Baseline, Week 12 (end of intervention)
  Plasma reduced glutathione measured by colorimetric assay and expressed in µmol/L. Higher values indicate better antioxidant status.
Oxidized Glutathione (GSSG, µmol/L) | Baseline, Week 12 (end of intervention)
  Plasma oxidized glutathione measured by colorimetric assay and expressed in µmol/L. Higher values indicate greater oxidative stress.
Thiobarbituric Acid Reactive Substances (TBARS, nmol MDA equivalents/mL plasma) | Baseline, Week 12 (end of intervention)
  Lipid peroxidation index measured as TBARS and expressed in nmol MDA equivalents/mL of plasma. Higher values indicate greater oxidative stress.
Malondialdehyde (MDA, µmol/L) | Baseline, Week 12 (end of intervention)
  Plasma MDA determined spectrophotometrically and expressed in µmol/L. Higher values indicate greater oxidative stress.
Total Antioxidant Capacity (TAC, mmol Trolox equivalents/L) | Baseline, Week 12 (end of intervention)
  Plasma TAC measured using colorimetric assay and expressed as mmol Trolox equivalents/L. Higher values indicate better antioxidant defense.
Relative expression levels of selected circulating microRNAs | Baseline, Week 12 (end of intervention), and 3-month follow-up
  Changes in the relative expression levels of selected circulating microRNAs associated with muscle metabolism, neuromuscular function, inflammation, oxidative stress, and anabolic signaling pathways. MicroRNAs will be quantified from peripheral blood samples using molecular profiling techniques.
Relative expression levels of selected exosome-derived microRNAs | Baseline and Week 12
  Changes in the relative expression levels of selected exosome-derived microRNAs related to muscle function, inflammation, and metabolic regulation, analyzed from circulating extracellular vesicles isolated from plasma samples.
Frequency of selected genetic variants related to creatine and HMB responsiveness | Baseline
  Analysis of the frequency of selected genetic variants related to muscle metabolism, anabolic signaling, and exercise responsiveness to explore interindividual variability in functional and molecular responses to creatine and HMB supplementation.
Relative abundance of selected circulating proteins involved in muscle and inflammatory responses | Baseline and Week 12
  Changes in the relative abundance of selected circulating proteins involved in muscle metabolism, inflammation, oxidative stress, and functional adaptation in response to creatine and HMB supplementation combined with exercise. Protein abundance will be assessed using targeted proteomic approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Mielgo-Ayuso, PhD, Study Chair — Universidad de Burgos
Locations (1):
- Residencia de Mayores Fuentes Blancas (Diputación Provincial de Burgos), Burgos, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results of this trial (including baseline characteristics and outcome measures) will be made available to qualified researchers upon reasonable request. Data will be shared only after publication of the main results and following approval of a research proposal and data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 6 months after publication of the main results, for at least 5 years.
Access Criteria: Researchers may request access by contacting the Principal Investigator (Prof. Juan Mielgo-Ayuso, Universidad de Burgos). Requests will be reviewed by the study steering committee. Access will be granted to qualified researchers whose proposals are scientifically and ethically sound, and who agree to sign a data access agreement.

REFERENCES:
- [Result] Rezola-Pardo C, Rodriguez-Larrad A, Gomez-Diaz J, Lozano-Real G, Mugica-Errazquin I, Patino MJ, Bidaurrazaga-Letona I, Irazusta J, Gil SM. Comparison Between Multicomponent Exercise and Walking Interventions in Long-Term Nursing Homes: A Randomized Controlled Trial. Gerontologist. 2020 Sep 15;60(7):1364-1373. doi: 10.1093/geront/gnz177. PMID 31845733
- [Result] Fernandez-Landa J, Calleja-Gonzalez J, Leon-Guereno P, Caballero-Garcia A, Cordova A, Mielgo-Ayuso J. Effect of the Combination of Creatine Monohydrate Plus HMB Supplementation on Sports Performance, Body Composition, Markers of Muscle Damage and Hormone Status: A Systematic Review. Nutrients. 2019 Oct 20;11(10):2528. doi: 10.3390/nu11102528. PMID 31635165
- [Result] Fernandez-Landa J, Fernandez-Lazaro D, Calleja-Gonzalez J, Caballero-Garcia A, Cordova A, Leon-Guereno P, Mielgo-Ayuso J. Long-Term Effect of Combination of Creatine Monohydrate Plus beta-Hydroxy beta-Methylbutyrate (HMB) on Exercise-Induced Muscle Damage and Anabolic/Catabolic Hormones in Elite Male Endurance Athletes. Biomolecules. 2020 Jan 15;10(1):140. doi: 10.3390/biom10010140. PMID 31952174
- [Result] Fernandez-Landa J, Fernandez-Lazaro D, Calleja-Gonzalez J, Caballero-Garcia A, Cordova Martinez A, Leon-Guereno P, Mielgo-Ayuso J. Effect of Ten Weeks of Creatine Monohydrate Plus HMB Supplementation on Athletic Performance Tests in Elite Male Endurance Athletes. Nutrients. 2020 Jan 10;12(1):193. doi: 10.3390/nu12010193. PMID 31936727
- [Result] Holecek M. Beta-hydroxy-beta-methylbutyrate supplementation and skeletal muscle in healthy and muscle-wasting conditions. J Cachexia Sarcopenia Muscle. 2017 Aug;8(4):529-541. doi: 10.1002/jcsm.12208. Epub 2017 May 10. PMID 28493406
- [Result] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Result] Devries MC, Phillips SM. Creatine supplementation during resistance training in older adults-a meta-analysis. Med Sci Sports Exerc. 2014 Jun;46(6):1194-203. doi: 10.1249/MSS.0000000000000220. PMID 24576864
- [Result] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372